CLINICAL TRIAL: NCT00959803
Title: An Investigator- And Subject-Blind Phase 1 Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of PF-04447943 After Administration Of Single Oral Doses To Healthy Young Adult Japanese Subjects And Multiple Oral Doses To Healthy Elderly Japanese Subjects
Brief Title: Study Of Single Ascending And Multiple Doses Of PF-04447943 In Japanese Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B0401004
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Phase 1; Pharmacokinetics; Healthy Young Adult; Japanese; Healthy Elderly; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose (Experimental): 3 way crossover with randomized placebo substitution to evaluate single escalating oral doses of PF 04447943 in 9 healthy young adult subjects.
  Interventions: Drug: PF-04447943; Drug: Placebo
- Multiple dose (Experimental): 3:1 active PF 04447943 to placebo randomization in 8 healthy elderly subjects.
  Interventions: Drug: PF-04447943; Drug: Placebo

INTERVENTIONS:
Drug: PF-04447943 — 3 mg solution, oral single dose.
  Arms: Single dose
Drug: PF-04447943 — 10 mg solution, oral single dose.
  Arms: Single dose
Drug: PF-04447943 — 25 mg solution, oral single dose.
  Arms: Single dose
Drug: Placebo — Solution, oral single dose.
  Arms: Single dose
Drug: PF-04447943 — 25 mg solution, oral twice daily for 7 days.
  Arms: Multiple dose
Drug: Placebo — Solution, oral twice daily for 7 days.
  Arms: Multiple dose

SUMMARY:
This study is designed to investigate the safety, tolerability, and pharmacokinetics of PF-04447943 after single and multiple-dose administration to healthy young adult and elderly Japanese subjects, respectively.

ELIGIBILITY:
Inclusion Criteria:

* For young cohort, healthy male and/or female Japanese of non-child bearing potential between the age of 18 and 55 years, inclusive.
* For elderly cohort, healthy male and/or female Japanese of non-child bearing potential between the age of 65 and 85 years, inclusive.
* Body Mass Index (BMI) between 17.5 to 30.5 kg/m2, and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Pregnant or nursing women; women of childbearing potential.
* Males who are unwilling to abstain from sexual intercourse or use a condom with all child-bearing potential women for the duration of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
AEs (spontaneous and solicited). Change from baseline in vital signs. | Day 0 to follow up visit after Study Day 5(single dose arm) and Day 11(multiple dose arm)
ECG and clinical safety laboratory endpoints, including a complete blood count, a full chemistry panel (including electrolytes and hepatic transaminases) and urinalysis. | Screening visit to follow up visit after Study Day 5(single dose arm) and Day 11(multiple dose arm)
Pharmacokinetic (single): AUClast, Cmax, Tmax | Day 1 to day 5
Pharmacokinetic(multiple): AUCt, Cmax and Tmax on Days 1 and 7, and Ctrough on Days 2, 3, 4 and 7. | Day 1 to day 11

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401004&StudyName=Study%20Of%20Single%20Ascending%20And%20Multiple%20Doses%20Of%20PF-04447943%20In%20Japanese%20Subjects.